CLINICAL TRIAL: NCT05301465
Title: Prospective Study to Identify and Validate the Predictive Role of Circulating Angiogenic Factors in Patients With Metastatic Gastric Cancer Treated With Second-line Paclitaxel and Ramucirumab
Brief Title: Predictive Role of Circulating Angiogenic Factors for Second-line Paclitaxel and Ramucirumab.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Gianluca Masi, Associate Professor, University of Pisa
Other Study IDs: PREDICTOR
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer Stage IV
Keywords: ramucirumab; gastric cancer; paclitaxel; predictive factors; VEGF
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project is primarily aimed at identifying and subsequently validating the predictive role of plasma concentrations of VEGF-A (vascular endothelial growth factor A), VEGF-D (vascular endothelial growth factor D) and s-VEGFR2 (soluble Vascular Endothelial Growth Factor Receptor 2) measured prior to initiation and during second-line treatment with paclitaxel and ramucirumab in patients with unresectable gastric cancer pretreated with first-line chemotherapy.

For the primary endpoint, the efficacy parameter chosen is PFS, calculated from day 1 of treatment to date of progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the stomach, cardia or gastroesophageal junction;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1;
* Life expectancy >3 months;
* Age >18 years;
* Metastatic disease measurable or evaluable according to RECIST (Response Evaluation Criteria in Solid Tumors) 1.1;
* Progression after previous first-line treatment with fluoropyrimidines and platinum derivative; previous neoadjuvant/adjuvant treatment terminated ≤6 months after instrumental evidence of relapse will be considered first-line treatment;
* Prior treatment with trastuzumab in case of HER-2 (human epidermal growth factor receptor 2) positive disease, defined as a 3+ immunohistochemistry (IHC) or 2+ IHC score and subsequent gene amplification demonstrated by Fluorescent In Situ Hybridization (FISH);

Exclusion Criteria:

* Previous treatment with ≥2 lines of systemic therapy for metastatic disease;
* Symptomatic peripheral neuropathy ≥2 grades according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03;
* Uncontrolled infections in active phase, disseminated intravascular coagulation in activity;
* Clinically significant cardiovascular disease, such as cardiovascular accidents (less than 6 months after initiation of treatment), myocardial infarction (less than 6 months after initiation of treatment), unstable angina, chronic heart failure ≥2 New York Heart Association (NYHA) grade, uncontrolled arrhythmias;
* Past (within 2 years of treatment initiation, except for curatively treated basal or squamous cell carcinomas of the skin or carcinoma in situ of the cervix) or current history of malignancy other than gastric cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled are affected by metastatic gastro-oesophageal junction or stomach cancer, undergoing second-line treatment with the combination of paclitaxel and ramucirumab according to normal clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | PFS is defined as the time interval between the start of second-line treatment and documentation of disease progression or death (whichever occurs first), assessed up to 6 months for each enrolled patient.
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided